CLINICAL TRIAL: NCT02465645
Title: A Prospective Randomized Study to Compare the Efficacy and Safety of Carvedilol With or Without Simvastatin in Patients With Portal Hypertension and Esophageal Varices
Brief Title: To Compare the Efficacy and Safety of Carvedilol With or Without Simvastatin in Patients With Portal Hypertension and Esophageal Varices.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-004
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2017-01

CONDITIONS: Cirrhosis With Esophageal Varices
MeSH Terms: interventions — Carvedilol; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol + Simvastatin (Experimental): Carvedilol will be administered orally at a start dose of 3.125 mg twice daily per day. After 1 week, this will increased to a dose of 6.25 mg twice daily per day. Target dose of 12.5 mg twice daily per day will be started after 2 weeks if systolic blood pressure does not fall below 90 mm Hg and HR 55-60/min.
  Simvastatin will be administered orally at a start dose of 20 mg for 15 days followed by 40 mg OD for the next 3 months. Along with Simvastatin, Carvedilol will be administered orally at a start dose of 3.125 mg twice daily per day. After 1 week, this will increased to a dose of 6.25 mg twice daily per day. Target dose of 12.5 mg twice daily per day will be started after 2 weeks if systolic blood pressure does not fall below 90 mm Hg and HR 55-60/min.
  Interventions: Drug: Carvedilol + Simvastatin
- Carvedilol (Active Comparator): Carvedilol will be administered orally at a start dose of 3.125 mg twice daily per day. After 1 week, this will increased to a dose of 6.25 mg twice daily per day. Target dose of 12.5 mg twice daily per day will be started after 2 weeks if systolic blood pressure does not fall below 90 mm Hg and HR 55-60/min.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol
  Arms: Carvedilol
Drug: Carvedilol + Simvastatin
  Arms: Carvedilol + Simvastatin

SUMMARY:
After successful screening of patients based on inclusion criteria, we will measure the baseline Hepatic Venous Pressure Gradient. At day 1 patients will undergo complete blood investigation including complete haemogram, kidney function test, liver function test, prothrombin time, AFP (Alfa Feto Protein) level, chest x ray, ultrasonography, fibroscan. Routine complete physical examination will be done.

ELIGIBILITY:
Inclusion Criteria:

1. All patients of chronic liver disease with esophageal varices.
2. Age more than and equal to 18 years.

Exclusion Criteria:

1. Patients of chronic liver disease with history of upper Gastro Intestinal bleed.
2. Patients of acute on chronic liver failure
3. Thrombosis of splenoportal axis
4. Hepatocellular carcinoma
5. Patients who were on primary variceal ligation sessions as prophylaxis
6. Patients who are beta blocker intolerant (Prior h/o hypotension, bradycardia).
7. Patients who are contraindicated for beta blockers {H/O COPD (Coronary Obstructive Pulmonary Disease), heart block, refractory Ascites, SBP(Spontaneous Bacterial Peritonitis) , HRS(Hepato Renal Syndrome)}.
8. Failure to give consent for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Total number of patients who will be Responders. | 3 Months
  Responders (Absolute value of HVPG<12 mm Hg or HVPG≥20% reduction)

SECONDARY OUTCOMES:
Total number of patients develop esophageal variceal bleed | 3 months
Total number of patients develop PHG (Portal Hypertensive Gastropathy). | 3 months
Total number of patients develop GAVE (Gastric Antral Vascular Ectasia). | 3 months
Total number of patients develop Gastric Varices. | 3 months
Total number of patients develop adverse Events of the study drug | 3 months
Improvement in the CTP (Child-Turcotte-Pugh score) score. | 3 months
Improvement in the MELD (Model for End Stage liver Disease) score. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr V Rajan, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Vijayaraghavan R, Jindal A, Arora V, Choudhary A, Kumar G, Sarin SK. Hemodynamic Effects of Adding Simvastatin to Carvedilol for Primary Prophylaxis of Variceal Bleeding: A Randomized Controlled Trial. Am J Gastroenterol. 2020 May;115(5):729-737. doi: 10.14309/ajg.0000000000000551. PMID 32079861